CLINICAL TRIAL: NCT00031174
Title: Collection Of Blood Components Using Apheresis From Patients With Rheumatic or Kidney Diseases and Healthy Volunteers
Brief Title: Blood Component Collection From Patients With Rheumatic or Kidney Disease and Healthy Volunteers
Status: Terminated | Type: Observational
Why Stopped: Due to technical and logistical constraints and a change in the study team's focus of research
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020131; 02-AR-0131
Record Dates: First submitted 2002-02-26; First posted 2002-02-27 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Rheumatic Diseases; Healthy Volunteers
Keywords: Apheresis; Healthy Volunteer; Rheumatoid Disease; Rheumatic Disease; Lupus; Rheumatoid Arthritis; Myositis; HV; Normal Control
MeSH Terms: conditions — Rheumatic Diseases; Arthritis, Rheumatoid; Myositis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Blood components collected using apheresis from normal volunteers.
- 2: Blood components collected using apheresis from patients with rheumatic or kidney diseases.

SUMMARY:
This study will collect white blood cells or plasma (the liquid part of the blood), or both, from healthy volunteers and from patients with rheumatic or kidney disorders for research purposes. Rheumatic disorders involve abnormalities of the immune system, the body s defense against disease. The immune system consists of white blood cells such as lymphocytes and monocytes, which produce substances such as antibodies and cytokines. White cells and plasma will be collected through a procedure called apheresis (described below).

Healthy volunteers and patients with confirmed or suspected rheumatic or kidney disease who are 18 years of age or older may be eligible for this study. Patients must be participating in a current protocol of the National Institute of Arthritis and Musculoskeletal and Skin Diseases or the National Institute of Digestive, Diabetes and Kidney Diseases. All candidates will be screened with a history, physical examination, and blood tests for hepatitis B and C and HIV infection. Women of childbearing age will be tested for pregnancy. Routine blood tests will be done in all volunteers, and in patients where needed. Pregnant women and people who test positive for hepatitis or HIV may not participate.

Participants will undergo apheresis to collect lymphocytes, monocytes, or plasma from the blood. For this procedure, a needle is placed in a vein in the arm. Blood flows from the vein through a tube (catheter) into a machine that spins the blood, separating it into its components. The required cells or plasma are extracted, and the rest of the blood, including the red cells and platelets, is returned to the body through the same needle or through a second needle placed in the other arm.

Cells collected from volunteers will be used in studies comparing the number and function of similar cells from patients with rheumatic diseases, focusing on the differences in number and function of the cells in health and disease. Components collected from patients will be used only for studies described in the protocol in which they are currently enrolled.

...

DETAILED DESCRIPTION:
Blood components will be collected using apheresis from normal volunteers and patients with rheumatic or kidney diseases. Mononuclear cells and plasma will be used by various investigators for research studies.

ELIGIBILITY:
* INCLUSION CRITERIA - Subjects with Rheumatic Diseases:

Patients with a diagnosed or suspected rheumatic or kidney disease, who are actively involved in a NIAMS or NIDDK protocol (have a current, signed consent form)

Ability to give informed consent

Age greater than or equal to 18 years

EXCLUSION CRITERIA - Subjects with Rheumatic Diseases:

History of allergy to acid-citrate-dextrose (ACD) anticoagulant

History of bleeding diatheses

Hemoglobin less than 9.0 g/dL

Platelet count less than 50,000/mm(3)

Pregnancy

Inadequate peripheral venous access

Active hepatitis B, C and/or HIV infection

Symptomatic coronary artery or valvular heart disease

Any concomitant illness that in the opinion of the investigators will substantially increase the risk of apheresis.

INCLUSION CRITERIA - Healthy Volunteers:

Subjects shall meet all donor eligibility criteria for autologous blood donation recommended or required by the Standards of the American Association of Blood Banks (1) and the Code of Federal Regulations of the Food and Drug Administration (2), with the exception of the travel exclusions related to malaria exposure and hypothetical exposure to the agent of variant Creutzfeldt-Jacob disease.

Ability to give informed consent

Age greater than or equal to 18 years

EXCLUSION CRITERIA - Healthy Volunteers:

History of autoimmune or chronic rheumatic disease within the last 5 years, with the exception of osteoarthritis

Active hepatitis B, C, and/or HIV infection

History of allergy to acid-citrate (ACD) anticoagulant

History of coagulopathies and bleeding diatheses

Symptomatic coronary artery disease or valvular heart disease

Hemoglobin less than 12.0 g/dL

Platelet count less than 100,000/cubic mm

Pregnancy

Inadequate peripheral venous access

Any concomitant illness that in the opinion of the investigators will substantially increase the risk of apheresis or make the volunteer ineligible for study controls are needed for (eg: active infection, allergies, etc.)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Rheumatic or kidney diseases and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2002-02-13 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
PBMC and Mononuclear cell study | 1/1/2030
  Blood components will be collected using apheresis from normal volunteers and patients with rheumatic or kidney diseases. Mononuclear cells and plasma will be used by various investigators for research studies.

CONTACTS AND LOCATIONS:
Overall Officials: Sarfaraz A Hasni, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2002-AR-0131.html